CLINICAL TRIAL: NCT01241097
Title: Comparison of the Effect on Endothelial Function of Statin Therapy in High Dose Versus Low Dose Combined With Ezetimibe
Brief Title: Pleiotropism of Statin Therapy in High Dose Versus Low Dose Combined With Ezetimibe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Bahia (Other)
Collaborators: Escola Bahiana de Medicina e Saude Publica (Other)
Responsible Party: Luis Claudio Lemos Correia, Phd, Escola Bahiana de Medicina e Saude Publica
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: sxse
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-06

CONDITIONS: Endothelial Function
Keywords: endothelial function; statins; ezetimibe; pleiotropism
MeSH Terms: interventions — Simvastatin; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- high-dose simvastatin, combined, placebo (Experimental): simvastatin 80 mg per days or simvastatin 10 mg and ezetimibe 10 mg, over a period of eight weeks, treatment consisted of tablets identical, or placebo
  Interventions: Drug: simvastatin, combined with simvastatin ezetimibe, placebo

INTERVENTIONS:
Drug: simvastatin, combined with simvastatin ezetimibe, placebo — simvastatin 80 mg per days or simvastatin 10 mg and ezetimibe 10 mg, over a period of eight weeks, treatment consisted of tablets identical, or placebo
  Other Names: zocor, vytorin

SUMMARY:
* To test the hypothesis that therapy with high dose statin provides endothelial superior benefit to the same cholesterol lowering with low-dose statin combined with ezetimibe.
* To test the hypothesis that therapy with high dose statin provides anti-inflammatory effect than the same reduction of cholesterol with low dose of statin plus ezetimibe

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled study. Inclusion Criteria: Obese women with body mass index (BMI)> 25 kg / m², aged 18 years and LDL-C> 100 mg / dl For treatment with simvastatin 80 mg, the participant will receive two identical vials, each containing a simvastatin 40 mg. For treatment with the combination simvastatin 10 mg and ezetimibe 10 mg, the participant will receive two identical bottles, one bottle with simvastatin 10 mg, and another bottle with ezetimibe 10mg. In the control group, each participant will receive two identical bottles, each bottle containing inert tablets. Each group with 20 participants.

Dependent Variable (Final Primary Outcome): Percentage change vasodilation of brachial artery flow-mediated, after treatment for eight weeks.

Covariates: clinical, biochemical markers and ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Women with body mass index (BMI)> 25 kg / m²
* Aged > 18 years
* LDL-C> 100 mg / dl

Exclusion Criteria:

* Previous use of statins, fibrates or ezetimibe
* Triglycerides> 400 mg / dl
* Serum creatinine greater than 2.0 md / dl
* Elevated liver enzymes, more than one and half times the upper limit of normal
* Creatine kinase (CK) levels more than three times the upper limit of normal
* Pregnant
* Breast-feeding
* Heart failure
* Psychiatric disorders
* Hormone replacement therapy.
* The occurrence of recent onset within the last four weeks of treatment with beta-blockers, converting enzyme inhibitor or calcium channel blocker, the intervention should be undertaken after a period of at least four weeks of continuous use.
* Acute inflammatory processes in the last month, assessed by clinical history and physical examination (ear, throat, skin lesions or other inflammatory manifestations) as well as reports of chronic diseases such as collagen, or the occurrence of active tuberculosis in the last three months will be excluded from work.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Percent change vasodilation of brachial artery flow-mediated, after eight weeks of treatment. | 8 weeks

SECONDARY OUTCOMES:
biochemical markers | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maristela M Garcia, MD, Principal Investigator — Escola Bahiana de Medicina e Saúde Pública
Locations (1):
- Escola Bahiana de Medicina e Saúde Púiblica, Salvador, Estado de Bahia, Brazil